CLINICAL TRIAL: NCT01197638
Title: Deutsches Ablations-Qualitätsregister
Brief Title: German Ablation Quality-Register
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: Ablations Register
Record Dates: First submitted 2010-07-29; First posted 2010-09-09 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Arrhythmia
Keywords: Cardiac arrhythmia; Catheter ablation; Register
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this register is the documentation of the success as well as of the complications regarding interventional therapy of cardiac arrhythmia by catheter ablation. This is the necessary basis for quality management and development of possible improvements of catheter ablation.

DETAILED DESCRIPTION:
The interventional therapy of heartbeat disturbances by means of catheter ablation makes the curative treatment possible of numerous tachycardiac arrhythmics. By this crucial improvement of the supply of patients and its quality of life a genuine healing of a multiplicity of heartbeat disturbances became possible. Especially within the range of the ablation treatment there are relatively few con-trolled studies, which would give a broad collection of the results of the catheter ablation in the different indication areas.

Aim of the registry:

Documentation of indication, hospital course and complications during long term follow-up of patients with catheter ablation

Design:

Prospective, multicenter registry; FU-duration 12 months.

Duration:

Phase I: 2 years

Inclusion criteria:

Catheter ablation (intention to treat)

Exclusion criteria:

Missing declaration of consent

ELIGIBILITY:
Inclusion Criteria:

* The ablation register will include all consecutive patients with a performed or attempted electrophysiological ablation

Exclusion Criteria:

* Missing signed informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consecutive patients with an performed or attempted electrophysiological ablation
Sampling Method: Non-Probability Sample
Enrollment: 20663 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Characterize consecutive patients with electrophysiological ablation in daily hospital routine in Germany. | 01/06/2008-12/31/2011

SECONDARY OUTCOMES:
Documentation of the technical implementation of ablation and the success of the intervention | 01/06/2008-12/31/2011
Documentation of further necessary interventions after the initial ablation during hospital stay | 01/06/2008-12/31/2011
Documentation of hospital mortality, serious but non-fatal complications (stroke, TIA, myocardial infarction, resuscitation), and complications caused by bleedings (serious as well as moderate) | 01/06/2008-12/31/2011
Documentation of medication therapy at hospital discharge | 01/06/2008-12/31/2011
Documentation of the 1-year mortality, serious but non-fatal complications (stroke, TIA, myocardial infarction, resuscitation), of heavy bleedings, of phrenicus pareses, PV-stenoses, or fistulas | 01/06/2008-12/31/2011
Documentation of the absence of relapse and of symptomatology after one year | 01/06/2008-12/31/2011
Documentation of needed interventions (implantation of either pacemaker, ICD or CRT, revascularization, a further ablation) during the first year after ablation | 01/06/2008-12/31/2011
Documentation of hospitalizations during the first year after ablation | 01/06/2008-12/31/2011
Documentation of medication therapy after 12 months | 01/06/2008-12/31/2011

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Senges, MD, Principal Investigator — Stiftung Institut fuer Herzinfarktforschung
Locations (9):
- Germany (9):
  - Herz- und Gefäßklinik, Bad Neustadt / Saale
  - Vivantes Klinikum Am Urban, Berlin
  - St. Marien Hospital, Bonn
  - Klinikum Coburg, Coburg
  - Praxisklinik Herz und Gefäß,, Dresden
  - Asklepios Klinik St Georg, Hamburg
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Städt Klinikum Hildesheim, Hildesheim
  - Krankenhaus München Bogenhausen, München

IPD SHARING:
Plan to Share IPD: No
Not included in informed consent.

REFERENCES:
- [Derived] Schleberger R, Metzner A, Kuck KH, Andresen D, Willems S, Hoffmann E, Deneke T, Eckardt L, Brachmann J, Hochadel M, Senges J, Rillig A. Antiarrhythmic drug therapy after catheter ablation for atrial fibrillation-Insights from the German Ablation Registry. Pharmacol Res Perspect. 2021 Dec;9(6):e00880. doi: 10.1002/prp2.880. PMID 34664789
- [Derived] Dechering DG, Gonska BD, Brachmann J, Lewalter T, Kuck KH, Andresen D, Willems S, Spitzer SG, Straube F, Schumacher B, Hochadel M, Senges J, Eckardt L. Efficacy and complications of cavo-tricuspid isthmus-dependent atrial flutter ablation in patients with and without structural heart disease: results from the German Ablation Registry. J Interv Card Electrophysiol. 2021 Jun;61(1):55-62. doi: 10.1007/s10840-020-00769-z. Epub 2020 May 27. PMID 32458180